CLINICAL TRIAL: NCT01613222
Title: SpO2 System Accuracy Testing
Brief Title: SpO2 System Accuracy Testing With Different Sensors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 118.02-2011-GES-0012
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Pulse Oximetry
MeSH Terms: interventions — Oximetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulse oximetry monitoring (Experimental): The U-TruSignal with different sensors is feasible for noninvasive and continuous SpO2 monitoring and meets the specified measurement accuracy when compared to a co-oximetry gold reference.
  Interventions: Device: Pulse oximetry

INTERVENTIONS:
Device: Pulse oximetry — Pulse oximetry measurement using SpO2 sensors, patient monitors, co-oximeters, and various modules.

SUMMARY:
A study to test the accuracy of SpO2 sensors with various patient monitors, co-oximeters, and modules.

DETAILED DESCRIPTION:
The U-TruSignal with different sensors is feasible for noninvasive and continuous SpO2 monitoring and meets the specified measurement accuracy when compared to a co-oximetry gold reference.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent or have a legally authorized representative provide written informed consent
* Subjects who are 18-55 years of age
* Subjects must be willing and able to comply with study procedures
* HbCO<3% (for smokers only)

Exclusion Criteria:

* Subject or a legally authorized representative is unable to provide written inform consent.
* Subjects that are considered morbidly obese (defined as BMI > 39.5),
* Subjects with injuries, deformities or abnormalities that may prevent proper application of the device under test,
* Smokers with COHb levels >3% or subjects who have smoked within two (2) days. Subjects will be screened for COHb levels of >3% with a Masimo Radical 7 (Rainbow).
* Subjects with known respiratory conditions (uncontrolled asthma, head cold, flu, pneumonia / bronchitis, respiratory distress / respiratory or lung surgery, emphysema, COPD, lung disease),
* Subjects with known heart or cardiovascular conditions,
* Female subjects that are actively trying to get pregnant or are pregnant,
* Subjects taking blood thinners or medications with aspirin or other antiplatelet medication in them (applies only to arterial draw study),
* Subjects with Systolic blood pressure >140mmHg,
* Subjects with Diastolic blood pressure >100mmHg,
* Subjects with heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2012-06-19 (Actual); Primary Completion 2013-02-15 (Actual); Study Completion 2013-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Conner, Study Director — GEHC
Locations (1):
- Clinimark, Louisville, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on June19, 2012 and the last subject was enrolled on February 15, 2013. The study was conducted at Clinimark, a human performance laboratory that tests physiological monitoring devices.
Groups:
- Pulse Oximetry Monitoring: Pulse oximetry : Pulse oximetry measurement using SpO2 sensors, patient monitors, co-oximeters, and various modules.
Period: Overall Study
Arm/Group | Pulse Oximetry Monitoring
Started | 63
Completed | 51
Not Completed | 12
Not completed — Physician Decision | 1
Not completed — Unable to place arterial line | 1
Not completed — Reused disposable sensors | 10

BASELINE CHARACTERISTICS:
Population: 63 subjects were enrolled. Data from 51 subjects was used for analysis.
Groups:
- Pulse Oximetry Monitoring: Pulse Oximetry Monitoring Single Arm
Arm/Group | Pulse Oximetry Monitoring
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.4 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 51
SpO2 [Mean (Standard Deviation); unit: % oxygen] | 95.1 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Accuracy Root Mean Square (ARMS)
Description: The Accuracy Root Mean Square (ARMS) calculation is used to measure accuracy of the test SpO2 device compared to reference SpO2 device. A scatterplot is created with the forehead sensor saturation on the y-axis and the measured blood saturation on the x-axis. The line of identity is drawn representing the ideal points, meaning that the forehead sensor saturation is always the same as the blood saturation. The dispersion of the actual data points around the line of identity can be measured using a statistical calculation called Arithmetic Root Mean Square (ARMS). The smaller ARMs the closer the data points lie around the line of identity, representing a more accurate sensor as accurate and appropriate. Data analysis follows ISO 80601-2-61, 2011, Annex EE and the FDA Guidance Document for Pulse Oximeters (FDA Draft Guidance, July 19, 2007).
Time Frame: 60 minutes
Population: The data analyzed was SpO2 data pairs using different U-Trusginal SpO2 sensors, patient monitors, co-oximeters, and various modules. Multiple data pairs were collected from each study participant, but not all sensors, patient monitors, co-oximeters and module configurations were used with each participant.
Measure: Mean (Full Range); unit: Accuracy Root Mean Square
Units Other Than Participants: Number of Data Pairs
Groups:
- Pulse Oximetry Monitoring Using SpO@ Sensors: Pulse oximetry measurement using different U-Trusginal SpO2 sensors, patient monitors, co-oximeters, and various modules.
Arm/Group | Pulse Oximetry Monitoring Using SpO@ Sensors
Number analyzed (Participants) | 51
Number analyzed (Number of Data Pairs) | 2826
Accuracy Root Mean Square
  TS-AAW Sensor + B40 Patient Monitor: number analyzed (Participants) | 10
  TS-AAW Sensor + B40 Patient Monitor: number analyzed (Number of Data Pairs) | 217
  TS-AAW Sensor + B40 Patient Monitor | 1.488 [-3.875 to 4.55]
  TS-AAW Sensor + 3900 Oximeter: number analyzed (Participants) | 10
  TS-AAW Sensor + 3900 Oximeter | 1.465 [-4.58 to 4.41]
  TS-AAW Sensor + Carescape V100 & UTrusignal V2: number analyzed (Participants) | 11
  TS-AAW Sensor + Carescape V100 & UTrusignal V2 | 1.651 [-3.5 to 7.1]
  TS-AAW Sensor + Carescape V100: number analyzed (Participants) | 11
  TS-AAW Sensor + Carescape V100 | 1.352 [-5.175 to 5]
  TS-AAW Sensor + EPRESTN: number analyzed (Participants) | 11
  TS-AAW Sensor + EPRESTN | 2.179 [-7.005 to 8.42]
  TS-AAW Sensor + M-NESTPR: number analyzed (Participants) | 10
  TS-AAW Sensor + M-NESTPR | 1.813 [-7.7 to 3.65]
  TS-AAW Sensor + M-OSAT: number analyzed (Participants) | 10
  TS-AAW Sensor + M-OSAT | 1.496 [-2.9 to 4.55]
  TS-AAW Sensor + TruSat: number analyzed (Participants) | 11
  TS-AAW Sensor + TruSat | 1.612 [-4.865 to 7.71]
  TS-SA-D Sensor + TruSat: number analyzed (Participants) | 11
  TS-SA-D Sensor + TruSat | 1.523 [-3.65 to 7.07]
  TS-AAW Sensor + TruffSat: number analyzed (Participants) | 10
  TS-AAW Sensor + TruffSat: number analyzed (Number of Data Pairs) | 217
  TS-AAW Sensor + TruffSat | 1.286 [-3.275 to 4.55]

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- TS-AAW Sensor + 3900 Oximeter; TS-AAW Sensor + B40 Patient Monitor; TS-AAW Sensor + Carescape V100 With TruSignal V2 SpO2 Board; TS-AAW Sensor + Carescape V100; TS-AAW Sensor + EPRESTN; TS-AAW Sensor + M-NESTPR; TS-AAW Sensor + M-OSAT; TS-AAW Sensor + TruSat; TS-AAW Sensor + TuffSat; TS-SA-D Sensor + Carescape V100 With TruSignal V2 SpO2 Board: Pulse oximetry : Pulse oximetry measurement using SpO2 sensors, patient monitors, co-oximeters, and various modules.
Arm/Group | TS-AAW Sensor + 3900 Oximeter | TS-AAW Sensor + B40 Patient Monitor | TS-AAW Sensor + Carescape V100 With TruSignal V2 SpO2 Board | TS-AAW Sensor + Carescape V100 | TS-AAW Sensor + EPRESTN | TS-AAW Sensor + M-NESTPR | TS-AAW Sensor + M-OSAT | TS-AAW Sensor + TruSat | TS-AAW Sensor + TuffSat | TS-SA-D Sensor + Carescape V100 With TruSignal V2 SpO2 Board
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor cannot require changes to the PI's disclosure, with the exception of requesting the removal of sponsor's confidential information. The study results themselves are not considered confidential information. Sponsor cannot extend the embargo beyond 60 days unless the PI's disclosure contains patentable subject matter, in which an embargo beyond 60 days may be necessary to allow for the filing of a patent application